CLINICAL TRIAL: NCT00003834
Title: A Phase II Study of Patients With Unresectable Metastatic Adenocarcinoma of the Colon or Rectum (Per 04/99 Amendment) Old Title: A Phase II Study of Patients With Unresectable Metastatic Adenocarcinoma of the Colon or Rectum Confined to the Liver
Brief Title: Combination Chemotherapy in Treating Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-974651; CDR0000066991 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oxaliplatin + leucovorin + fluorouracil (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1, then leucovorin calcium IV over 2 hours with fluorouracil IV bolus, followed by fluorouracil IV over 22 hours on days 1 and 2. Courses repeat every 2 weeks. Patients with stable disease continue treatment in the absence of disease progression or unacceptable toxicity or until disease is resectable. Patients who achieve complete response (CR), partial response (PR) with unresectable disease, or PR but are not surgical candidates continue treatment in the absence of disease progression or unacceptable toxicity. Patients who demonstrate a response are treated until best response or until disease is deemed resectable. Patients who achieve a CR or PR and are resected may receive 2 to 4 additional courses of therapy at the discretion of the investigator. Patients are followed every 3 months for 1 year and then every 6 months for 2 years.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of treatment with oxaliplatin, fluorouracil, and leucovorin calcium in terms of the resectability rate in patients with unresectable advanced colorectal carcinoma confined to the liver. II. Assess this regimen in terms of response rate, toxicity, and overall survival in these patients.

OUTLINE: Patients receive oxaliplatin IV over 2 hours on day 1, then leucovorin calcium IV over 2 hours with fluorouracil IV bolus, followed by fluorouracil IV over 22 hours on days 1 and 2. Courses repeat every 2 weeks. Patients with stable disease continue treatment in the absence of disease progression or unacceptable toxicity or until disease is resectable. Patients who achieve complete response (CR), partial response (PR) with unresectable disease, or PR but are not surgical candidates continue treatment in the absence of disease progression or unacceptable toxicity. Patients who demonstrate a response are treated until best response or until disease is deemed resectable. Patients who achieve a CR or PR and are resected may receive 2 to 4 additional courses of therapy at the discretion of the investigator. Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: History of carcinoma of the colon or rectum in which the primary site has been completely resected Measurable or evaluable unresectable liver metastases with one or more of the following: Involvement of all 3 major hepatic veins, the portal vein bifurcation, or the retrohepatic vena cava Involvement of the main right or the main left portal vein and the main hepatic vein of the opposite lobe Disease requiring more than a right or left trisegmentectomy Six or more metastatic lesions distributed diffusely in both lobes of the liver

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT no greater than 3 times upper limit of normal (ULN) No chronic hepatic disease (e.g., chronic active hepatitis, cirrhosis) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No history of myocardial infarction within the past 6 months No congestive heart failure Other: No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of any organ or other tumor associated with less than 10% probability of death from malignant disease within 5 years of diagnosis Adequate oral nutrition including estimated intake of at least 1,500 calories per day No severe anorexia or frequent nausea and/or vomiting Able to withstand a major operative procedure No neuropathy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Concurrent filgrastim or epoetin alfa allowed Chemotherapy: At least one year since prior adjuvant systemic fluorouracil with or without levamisole or leucovorin No prior systemic or hepatic artery infusion chemotherapy for metastatic disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the liver At least one year since radiotherapy to greater than 25% of bone marrow No concurrent radiotherapy Surgery: At least 21 days since abdominal exploration with or without intestinal resection Other: Oral cryotherapy allowed only on day 2 of each course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 1999-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 4 years

SECONDARY OUTCOMES:
overall survival | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Alberts SR, Horvath WL, Sternfeld WC, Goldberg RM, Mahoney MR, Dakhil SR, Levitt R, Rowland K, Nair S, Sargent DJ, Donohue JH. Oxaliplatin, fluorouracil, and leucovorin for patients with unresectable liver-only metastases from colorectal cancer: a North Central Cancer Treatment Group phase II study. J Clin Oncol. 2005 Dec 20;23(36):9243-9. doi: 10.1200/JCO.2005.07.740. Epub 2005 Oct 17. PMID 16230673
- [Result] Alberts SR, Horvath W, Donohue J, et al.: Oxaliplatin (OXAL), 5-Fluorouracil (5FU), and Leucovorin (CF) for patients (Pts) with liver only metastases (Mets) from colorectal cancer (CRC): a North Central Cancer Treatment Group (NCCTG) phase II study. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-511, 2001.